CLINICAL TRIAL: NCT05251090
Title: A Phase I, Multicentre, Open-label Study to Evaluate the Safety and Pharmacokinetic of Recombinant Human Coagulation Factor VIII, Fc Fusion Protein for Injection in Children With Severe Hemophilia A
Brief Title: A Study to Evaluate the Safety and Pharmacokinetic of Recombinant Human Coagulation Factor VIII ，Fc Fusion Protein for Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Gensciences lnc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTR20220279
Record Dates: First submitted 2022-02-11; First posted 2022-02-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Hemophilia A
Keywords: Hemophilia A;Pharmacokinetics;Child;Safety and Tolerability
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Subjects(up to 12 years of age) received two treatments: 50 IU/kg ADVATE in the first period, followed by 50 IU/kg FRSW107 in the second period.
  Interventions: Drug: ADVATE; Drug: FRSW107

INTERVENTIONS:
Drug: ADVATE — 50 international units (IU)/kg, a single dose.
Drug: FRSW107 — 50 IU/kg, a single dose.
  Other Names: Recombinant Human Coagulation Factor VIII, Fc Fusion Protein for Injection

SUMMARY:
Primary objective: To assess the pharmacokinetics of Recombinant Human Coagulation Factor VIII, Fc Fusion Protein for Injection (FRSW107) Secondary objectives: To assess Safety and Tolerability by monitoring FVIII recovery and adverse events in Severe Hemophilia A.

ELIGIBILITY:
Key Inclusion Criteria:

* The activity of the coagulation factor VIII (FVIII:C) < 1%. Less than 6 years old Patients previously treated with FVIII concentrate (s) for a minimum of 50 exposure days (EDs) prior to study entry. 6 years old to 12 years old Patients previously treated with FVIII concentrate (s) for a minimum of 150 exposure days (EDs) prior to study entry.
* Normal prothrombin time or INR < 1.3.
* Negative lupus anticoagulant.

Key Exclusion Criteria:

* Hypersensitive to any of the excipients of the test materials (e.g. allergic to murine or hamster origin heterologous proteins).
* History of hypersensitivity or anaphylaxis associated with any FVIII or II immunoglobulin administration.
* Current FVIII inhibitor-positive or history of FVIII inhibitor-positive.
* Other coagulation disorder(s) in addition to hemophilia A.
* Infusion of any products containing FVIII within 72 h prior to administration.
* Significant hepatic or renal impairment (ALT and AST > 2×ULN; serum bilirubin level > 2 × upper limit of normal (ULN), BUN > 2×ULN, Cr > 2.0 ULN).
* One or more clinically significant tests for Human Immunodeficiency Virus (HIV), Antisyphilitic spirulina (TPHA) and Hepatitis C Virus (HCV) Antibody.
* Patients who received any anticoagulant or antiplatelet therapy within one week prior screening or need to receive an anticoagulant or antiplatelet therapy during the period of clinical trials.
* Patients having major surgery or receiving blood or bood components transfusion within 4 weeks prior screening or having planned major surgery schedule during the study.
* Patients who previously participated in the other clinical trials within one month prior to administration.
* Any life-threatening disease or condition which, according to the investigator's judgment, could not benefit from the trial participation.
* Patient who is considered by the other investigators not suitable for clinical study.

Max Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Hemophilia A is an X-chromosome-linked recessive inherited bleeding disorder caused by a deficiency of coagulation factor VIII (FVIII).
Enrollment: 13 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2022-05-09 (Actual)

PRIMARY OUTCOMES:
Maximum measured concentration of FVIII:C (Cmax) | Pre-dose and post dose up to 8 days.
  Measured by aPTT Clotting Assay.
Time required for the concentration of the drug to reach half of its original value (T1/2) | Pre-dose and post dose up to 8 days
  Measured by aPTT Clotting Assay.
Area Under the Curve to Infinity (AUC) | Pre-dose and post dose up to 8 days.
  Measured by aPTT Clotting Assay.
The measure of the efficiency of the body to remove the drug and the unit is the volume of the plasma or blood cleared of drug per unit time (CL). | Pre-dose and post dose up to 8 days.
  Measured by aPTT Clotting Assay.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE V5.0. | Post dose up to 32 days.
  Adverse events related to Recombinant Human Coagulation Factor VIII-Fc fusion protein for Injection according to Common Terminology Criteria for Adverse Events (CTCAE) NCI.V5.0.
Development of Inhibitor | Pre-dose and post dose up to 32 days.
  Measured by the Nijmegen-Modified Bethesda Assay.

CONTACTS AND LOCATIONS:
Overall Officials: Runhui Wu, PhD, Principal Investigator — Beijing Children's Hospital; Xiaoling Wang, MA.Sc, Principal Investigator — Beijing Children's Hospital
Locations (6):
- China (6):
  - Beijing Children's Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Shenzhen Children's Hospita, Shenzhen, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangzhou
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Chengdu Women's and Children's Central Hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No